CLINICAL TRIAL: NCT01195766
Title: Phase II-study Using Ofatumumab and ESHAP Followed by Autologous Trasplant of Hemopoietic Precursors for the Treatment of Classic Hodgkin's Lymphoma on Relapse, Partial Response or Refractory to First Line Treatment
Brief Title: Study of Ofatumumab and ESHAP for the Treatment of Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O-ESHAP-LH-2009; 2009-016026-13 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin; Ofatumumab; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): Ofatumumab in addition to ESHAP therapy
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab in addition with ESHAP therapy
  Other Names: ARZERRA

SUMMARY:
The aim of this study is to analyze the efficacy of O-ESHAP treatment for Hodgkin's lymphome patients that have a first line chemotherapy treatment failure due to refractoriness, partial response or relapsed.

In the same way, mortality, global survival and free-progression survival after O-ESHAP treatment and TAPH will also analyzed.

DETAILED DESCRIPTION:
In addition to the above:

* To asses the complete response rate after O-ESHAP.
* To asses the toxicity of O-ESHAP regimen
* To asses the stem cells mobilization capacity of O-ESHAP regimen
* To evaluate the final results of the whole procedure (O-ESHAP followed by high-dose chemotherapy and ASCT): transplant-related mortality (TRM), overall survival (OS), and progression free survival (PFS)
* To investigate the correlation between the overall response and CD20 expression by tumoral cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed relapsed, partial response or refractory classical HL after first line chemotherapy. They will be included irrespective of CD20 expression on HRS cells. CD20 expression will be analyzed on all available biopsies and this data will be recorded for further evaluation.
* Age 18 to 65 years. Patient >65 and <70 years old with ECOG < 2 and absence of comorbidities will be included in the study if considered adequate by the investigator.
* Leucocytes > 3,0 x 109/L and platelets > 100 x 109/L.
* ECOG < 2.
* No major organ dysfunction.
* Written informed consent.
* HIV negative.
* No active hepatitis B or C infection.
* Availability of histological report of biopsy at diagnosis or at relapse and availability of biopsy to be revised by reference pathologists.
* Absence of other neoplasia, except basocellular tumor or carcinoma of the uterine cervix in situ.
* Contraception measures in fertile females.

Exclusion Criteria:

* Subjects who have current active hepatic or biliary disease
* presence of pathology that would contraindicate the administration of chemotherapy
* HIV positive
* Hepatitis B or C infection
* history of other malignancies in addition to those specified in the inclusion criteria
* informed consent not signed
* Pregnant and / or breast-feeding or reproductive capacity adults who do not use an effective method of birth control during study treatment and at least six months later. An effective method is that used at least one barrier mechanism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Analysis of the global response rate (complete responses + partial responses) after O-ESHAP treatment | 4 years follow-up

SECONDARY OUTCOMES:
To analyze the complete response rate after O-ESHAP treatment. Further secondary outcomes as described in study summary | 4 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Martínez, MD, Study Director — Hospital Clinic i provincial de Barcelona
Locations (14):
- Spain (14):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Pau, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Instituto Catalan de Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Carlos Haya, Málaga, Malaga
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital Morales Messeguer, Murcia, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Clinico de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital Clinico de Valencia, Valencia, Valencia
  - Hospital Rio Hortega, Valladolid, Valladolid